CLINICAL TRIAL: NCT02328157
Title: Combined 25-gauge Vitrectomy and Cataract Surgery With Toric Intraocular Lens With Idiopathic Epiretinal Membrane.
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Kagawa University (Other)
Responsible Party: Principal Investigator, Akitaka Tsujikawa, Professor and Chairman, Kagawa University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: H26-061
Record Dates: First submitted 2014-12-13; First posted 2014-12-31 (Estimated); Last update posted 2018-03-07 (Actual); Status verified 2018-03

CONDITIONS: Cataract; Epiretinal Membrane; Corneal Astigmatism
MeSH Terms: conditions — Cataract; Epiretinal Membrane; Astigmatism | interventions — Vitrectomy; Cataract Extraction

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Cataract with ERM and astigmatism (Experimental): Eyes that have cataract and ERM with a preoperative corneal cylinder of more than 0.75 diopter.
  Interventions: Device: Vitrectomy with cataract surgery and toric IOL; Device: Vitrectomy with cataract surgery and common IOL

INTERVENTIONS:
Device: Vitrectomy with cataract surgery and toric IOL
Device: Vitrectomy with cataract surgery and common IOL

SUMMARY:
Toric intraocular lens (IOL) is now widely used for the cataract surgery with preoperative corneal astigmatism.

Symptomatic epiretinal membrane (ERM) is often treated with 25-gauge transconjunctival sutureless vitrectomy, resulting in good visual recovery. So far, however, limited information is available on the the stability of axis rotation, astigmatism correction, and improvement in uncorrected distance visual acuity, using astigmatism-correcting IOL in a 25-gauge transconjunctival sutureless vitrectomy combined with cataract surgery. In the current study, eyes with a preoperative corneal cylinder of more than 0.75 diopter had a triple procedure for idiopathic ERM using a toric IOL. Outcome measures will be the amount of IOL axis rotation, uncorrected visual acuity, corrected distance visual acuity, and corneal and refractive astigmatism up to 6 months postoperatively. We are expecting to show that postoperative IOL axis stability is similar to that reported for cataract surgery alone in vitrectomy (triple procedure) for idiopathic ERM with a toric IOL.

ELIGIBILITY:
Inclusion Criteria:

* Preoperative corneal cylinder of more than 0.75 diopter
* Symptomatic idiopathic epiretinal membrane
* Symptomatic cataract

Exclusion Criteria:

* Severe media opacity other cataract
* Eyes with other retinal disease, such as diabetic retinopathy, retinal vein occlusion, rhegmatogenous retinal detachment

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2015-01; Primary Completion 2018-10 (Estimated); Study Completion 2018-10 (Estimated)

PRIMARY OUTCOMES:
The degree of IOL axis rotation from the end of surgery | Six months after the inplantation

CONTACTS AND LOCATIONS:
Overall Officials: AKITAKA TSUJIKAWA, MD, Principal Investigator — Kagawa Univerisity Faculty of Medicine
Locations (1):
- Kagawa University Faculty of Medicine, Hiragi, Kagawa-ken, Japan